CLINICAL TRIAL: NCT05000736
Title: Comparative Effectiveness of Palbociclib Plus Aromatase Inhibitor Versus Fulvestrant Alone as Initial Endocrine Therapy for HR+/HER2- Advanced Breast Cancer in Chinese Clinical Practice: a Real-world Study
Brief Title: Comparative Effectiveness of Palbociclib Plus AI Versus Fulvestrant for HR+/HER2- ABC
Acronym: CAPACITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-BC-086
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hormone Receptor Positive Advanced Breast Cancer
MeSH Terms: interventions — palbociclib; Aromatase Inhibitors; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- palbociclib + aromatase inhibitor: Adult patients with HR+/HER2- advanced breast cancer who received the initial endocrine therapy of palbociclib plus aromatase inhibitor at the Cancer Hospital Chinese Academy of Medical Sciences from August 1, 2018 to December 31, 2020.
  Interventions: Drug: palbociclib + aromatase inhibitor
- fulvestrant: Adult patients with HR+/HER2- advanced breast cancer who received the initial endocrine therapy of fulvestrant monotherapy at the Cancer Hospital Chinese Academy of Medical Sciences from August 1, 2018 to December 31, 2020.
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: palbociclib + aromatase inhibitor — palbociclib + aromatase inhibitor therapy
  Groups: palbociclib + aromatase inhibitor
Drug: fulvestrant — fulvestrant monotherapy
  Groups: fulvestrant

SUMMARY:
A retrospective cohort study conducted at the Cancer Hospital Chinese Academy of Medical Sciences to compare the effectiveness of palbociclib plus AI therapy and fulvestrant monotherapy as initial endocrine therapy in the patients with HR+/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
This study is designed to be a retrospective cohort study conducted at the Cancer Hospital Chinese Academy of Medical Sciences. The target populations of this study are patients with HR+/HER2- advanced breast cancer who received the initial endocrine therapy of palbociclib plus AI or fulvestrant monotherapy from August 1, 2018 to December 31, 2020. It is expected to enroll 600 subjects in this study. The subjects' data such as demographics and other baseline characteristics, medications, prognosis, will be collected retrospectively, and statistical analysis of data will be conducted to compare the effectiveness outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women ≥18 years old;
2. Diagnosed with locally advanced (stage IIIb/IIIc) or metastatic (stage IV) breast cancer;
3. The molecular classification is pathologically confirmed as HR+/HER2-;
4. Palbociclib plus AI or fulvestrant monotherapy as initial endocrine therapy for advanced breast cancer for at least 1 cycle;
5. The follow-up time should be not less than 3 months after the start of palbociclib plus AI therapy or fulvestrant monotherapy.

Exclusion Criteria:

1. Subjects who have previously received chemotherapy, other CDK4/6 inhibitors or other endocrine monotherapy for advanced breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HR+/HER2- advanced breast cancer who received the initial endocrine therapy of palbociclib plus AI or fulvestrant monotherapy at the Cancer Hospital Chinese Academy of Medical Sciences from August 1, 2018 to December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Real-world progression-free survival (rwPFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  It is defined as the time (months) from the start of palbociclib+AI or fulvestrant monotherapy to progressive disease or all-cause mortality. The progressive disease is determined by clinicians based on the results of clinical evaluation, laboratory tests, imaging or pathological examinations. Patients who have not died or have not experienced progressive disease will be censored at the beginning of next-line treatment or at the last visit during the study period.

SECONDARY OUTCOMES:
Overall survival | From date of index treatment until date of death from any acuse or date of end of study, whichever came first, assessed up to 36 months.
  It is defined as the time (months) from the start of palbociclib+AI or fulvestrant monotherapy to all-cause mortality. Patients who have not died are censored on the study deadline.
Real-world tumor response (rwTR) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 36 months.
  Real world ORR is defined as the proportion of patients with complete response (CR) or partial response (PR) reported by doctors among all patients with response data available.Real world CBR is defined as the proportion of patients who have reached CR, PR, or stable disease (SD) for at least 24 weeks reported by the doctors among all patients with response data available.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China